CLINICAL TRIAL: NCT03389607
Title: The Role of SCUBE-1 in Ischemia-reperfusion Injury in Patients With Knee Prosthesis
Brief Title: The Role of SCUBE-1 in Ischemia-reperfusion Injury
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: scube1
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Gonarthrosis; Diabetes
Keywords: SCUBE-1
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic: the patients must have diabetic disease
  Interventions: Diagnostic Test: spinal anesthesia
- control: the patients must not have diabetic
  Interventions: Diagnostic Test: spinal anesthesia

INTERVENTIONS:
Diagnostic Test: spinal anesthesia — before spinal anesthesia, before 5 min opening of tourniquet and 2 hr after operation SCUBE-1, MDA and TAC will measured from plasma

SUMMARY:
One consequence of tissue damage caused by tourniquet is ischemia-reperfusion injury. Short-term ischemia leads to vasodilatation and reactive hyperemia resulting in post-ischemic reperfusion microcirculation failure and tissue edema that extends from 30 minutes to 4 hours.

SCUBE-1 is a newly defined cell surface molecule. It emerges from many developing cells, including endothelium and platelets. Immunohistochemical demonstration of subendothelial matrix deposition in atherosclerosis in humans. We did not find any study that showed the post-ischemic regression of scube 1, which was shown to be significantly higher in ischemic events in the literature.

in this study is aimed to investigate the location / sensitivity of SCUBE-1 in diabetics and nondiabetics after application of regional anesthesia for ischemia-reperfusion injury induced by tourniquet application in knee prosthesis attempts in our aimed patients and compare this with other total antioxidant status (TAS) and MDA of ischemia-reperfusion parameters

DETAILED DESCRIPTION:
After being taken to the operation room, the patient will be divided into two groups as group D (diabetic) and group K (control) by standardized anesthesia monitoring with 5-lead electrocardiogram (ECG), peripheral oxygen saturation (SpO2) and noninvasive blood pressure measurements.

In both groups, spinal anesthesia will be applied in a lateral decubitus position using a 22 gauge Quincke spinal needle from the interspinal space as 0.5% heavy marcaine 10-12.5 mg 1 min. Atropine 0.5 mg and ephedrine 5 mg should be administered if bradycardia develops in both groups. The disease tourniquet will be applied after induction, in accordance with the literature, to be above 150 mmHg of the systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* knee replacement surgery
* using a pneumatic tourniquet

Exclusion Criteria:

* coronary artery disease
* renal disorders
* cognitive disorders
* bleeding diathesis
* who have passed general anesthesia
* anti-inflammatory drugs treatment
* abnormal HbA1c values

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-70
Study Population: the patients who will go to surgery for gonarthrosis disease
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
SCUBE-1 | before spinal anesthesia, before 5 min opening of tourniquet and 2 hr after operation
  mean level of SCUBE-1

SECONDARY OUTCOMES:
malondialdehyde (MDA) | before spinal anesthesia, before 5 min opening of tourniquet and 2 hr after operation
  mean level of MDA
total antioxidant capacity | before spinal anesthesia, before 5 min opening of tourniquet and 2 hr after operation
  mean level of total antioxidant capacity (TAC)

CONTACTS AND LOCATIONS:
Locations (1):
- university of health siences diskapi yildirim beyazit T&R hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No